CLINICAL TRIAL: NCT02006693
Title: Post Market Multicentric Evaluation of the AqueSys XEN Implant in Moderate Primary Open Angle Glaucoma Subjects
Brief Title: Evaluation of the XEN Implant in Moderate Primary Open Angle Glaucoma (POAG) Participants
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AqueSys, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MS-001
Record Dates: First submitted 2013-12-02; First posted 2013-12-10 (Estimated); Results first posted 2019-04-22 (Actual); Last update posted 2019-04-22 (Actual); Status verified 2019-01

CONDITIONS: Primary Open Angle Glaucoma
Keywords: XEN; Primary Open Angle Glaucoma; Filtration Device; Ab interno
MeSH Terms: conditions — Glaucoma, Open-Angle | interventions — Cataract Extraction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- XEN® Gel Stent (Other): The XEN®45 Gel Stent (XEN45 implant) was placed in the study eye as a standalone procedure.
  Interventions: Device: XEN® Gel Stent
- XEN® Gel Stent with Cataract Surgery (Other): The XEN® Gel Stent (XEN45 implant) with cataract surgery, occurred if the participant was diagnosed with a cataract.
  Interventions: Procedure: Cataract Surgery

INTERVENTIONS:
Device: XEN® Gel Stent — The XEN® Gel Stent (XEN45 implant) was placed in the study eye.
  Other Names: XEN Glaucoma Implant; XEN Gel Stent; XEN45 Implant
  Arms: XEN® Gel Stent
Procedure: Cataract Surgery — Participants diagnosed with a cataract elected to have cataract surgery.
  Arms: XEN® Gel Stent with Cataract Surgery

SUMMARY:
The objective of this study was to evaluate the AqueSys XEN Implant [XEN® Gel Stent (XEN45 Implant)] for the treatment of moderate primary open angle glaucoma (POAG) participants when medications have failed to control intraocular pressure (IOP). Effectiveness was evaluated by comparing medicated preoperative IOP to postoperative values. Additionally, the number of topical IOP-lowering medications at screening were compared to the number of IOP-lowering medications at 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of primary open angle glaucoma
* Participants are taking at least one and no more than four topical IOP-lowering medications.

Exclusion Criteria:

* Angle Closure Glaucoma
* Participant has neovascular, uveitic or angle recession glaucoma or any glaucoma associated with vascular disorders
* Clinically significant inflammation or infection in the study eye within 30 days prior to the preoperative visit (e.g., blepharitis, conjunctivitis, keratitis, uveitis, herpes simplex infection)
* Presence of conjunctival scarring or prior conjunctival surgery or other conjunctival pathologies (e.g., pterygium) in the target quadrant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 199 (Actual)
Dates: Start 2013-12-05 (Actual); Primary Completion 2016-02-09 (Actual); Study Completion 2017-01-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vanessa Vera, MD, Study Director — Allergan
Locations (21):
- Austria (3):
  - University of Graz, Graz
  - University Augenklinik Salzburg, Salzburg
  - Vienna University, Vienna
- University Hospitals Leuven, Leuven, Belgium
- Germany (3):
  - University Eye Clinic Bochum-Langendreer, Bochum
  - Klinik für Augenheilkunde, Frankfurt
  - Klinik fur Augenheilkunde, Neubrandenburg
- Italy (3):
  - University of Pisa, Pisa
  - Clinica Oculistica, Universita' di Torino, Torino
  - Integrated University Hospital of Verona, Verona
- Ophthalmology Department of the Military Health Service Institute, Warsaw, Poland
- Spain (3):
  - Hospital Meixeiro Servicio de Ofthalmologia, Vigo, Pontevedra
  - Hospital Universitario La Paz, Madrid
  - Hospital Principe de Asturias, Madrid
- University of Geneva, Geneva, Switzerland
- United Kingdom (5):
  - Maidstone Hospital Eye, Ear and Mouth Unit, Maidstone, Kent
  - Birmingham Midland Eye Theaters, Birmingham, West Midlands
  - Moorfields Eye Hospital, London
  - St. Thomas Hospital, London
  - Pinderfields Hospital, Wakefield
- Unidad Oftalmologica de Caracas, Caracas, Venezuela

REFERENCES:
- [Derived] Reitsamer H, Sng C, Vera V, Lenzhofer M, Barton K, Stalmans I; Apex Study Group. Two-year results of a multicenter study of the ab interno gelatin implant in medically uncontrolled primary open-angle glaucoma. Graefes Arch Clin Exp Ophthalmol. 2019 May;257(5):983-996. doi: 10.1007/s00417-019-04251-z. Epub 2019 Feb 13. PMID 30758653
- [Derived] Ozal SA, Kaplaner O, Basar BB, Guclu H, Ozal E. An innovation in glaucoma surgery: XEN45 gel stent implantation. Arq Bras Oftalmol. 2017 Nov-Dec;80(6):382-385. doi: 10.5935/0004-2749.20170093. PMID 29267575

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Eyes
Groups:
- XEN® Gel Stent: The XEN® Gel Stent (XEN45 implant) was placed in the study eye as a standalone procedure.
Period: Overall Study
Arm/Group | XEN® Gel Stent | XEN® Gel Stent With Cataract Surgery
Started | 112; 120 Eyes | 87; 98 Eyes
Completed | 84; 91 Eyes | 74; 83 Eyes
Not Completed | 28; 29 Eyes | 13; 15 Eyes
Not completed — No Reason Specified | 6 | 8
Not completed — Another Glaucoma-related Surgery | 12 | 1
Not completed — XEN Implant Explantation | 0 | 1
Not completed — Death | 2 | 2
Not completed — Lost to Follow-up | 4 | 1
Not completed — Patient Decision | 4 | 0

BASELINE CHARACTERISTICS:
Population: Modified Intent-to-Treat (mITT) Population included all eligible eyes that met IOP and IOP-lowering medication inclusion criteria and received the XEN45 implant.
Units Other Than Participants: Eyes
Groups:
- Total: Total of all reporting groups
Arm/Group | XEN® Gel Stent | XEN® Gel Stent With Cataract Surgery | Total
Number analyzed (Participants) | 106 | 79 | 185
Number analyzed (Eyes) | 114 | 88 | 202
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.3 (11.7) | 76.5 (6.1) | 71.8 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 55 | 40 | 95
  Male | 51 | 39 | 90
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 103 | 75 | 178
  Black or African American | 2 | 1 | 3
  Asian | 1 | 3 | 4

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Mean Intraocular Pressure (IOP) in the Study Eye to Month 12
Description: IOP is a measurement of the fluid pressure inside the eye. Two IOP measurements were taken, followed by a third if the first 2 differed by 3 mmHg or more. The measurements were averaged. The study eye(s) is defined as an eye(s) that met IOP and IOP-lowering medication study inclusion criteria. A negative change from Baseline indicates improvement.
Time Frame: Baseline (≤ 90 days Preoperative) to Month 12 (Postoperative)
Population: mITT Population included all eligible eyes that met IOP and IOP-lowering medication inclusion criteria and received the XEN45 implant. Number analyzed is the number of eyes with data at the given time-point.
Measure: Mean (Standard Deviation); unit: mmHg
Units Other Than Participants: eyes
Arm/Group | XEN® Gel Stent | XEN® Gel Stent With Cataract Surgery
Number analyzed (Participants) | 106 | 79
Number analyzed (eyes) | 114 | 88
mmHg
  Baseline (preoperation) | 21.7 (3.76) | 21.0 (3.39)
  Change from Baseline to Month 12: number analyzed (eyes) | 97 | 81
  Change from Baseline to Month 12 | -6.6 (5.64) | -6.4 (4.96)

2. Primary Outcome: Change From Baseline in the Number of Topical IOP-Lowering Medications in the Study Eyes to Month 12
Description: The use of topical IOP-lowering medications was recorded at the preoperative screening visit and at the 12 Month postoperative visit. The study eye(s) is defined as an eye(s) that met IOP and IOP-lowering medication study inclusion criteria. A negative change from Baseline indicates improvement.
Time Frame: Baseline (≤ 90 days Preoperative) to Month 12 (Postoperative)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: medications
Units Other Than Participants: eyes
Arm/Group | XEN® Gel Stent | XEN® Gel Stent With Cataract Surgery
Number analyzed (Participants) | 106 | 79
Number analyzed (eyes) | 114 | 88
medications
  Baseline (preoperation) | 2.7 (0.93) | 2.5 (0.88)
  Change from Baseline to Month 12: number analyzed (eyes) | 97 | 81
  Change from Baseline to Month 12 | -1.8 (1.31) | -1.6 (1.17)

3. Primary Outcome: Mean Change From Baseline in IOP in the Study Eyes to Month 24
Description: as for outcome 1
Time Frame: Baseline (≤ 90 days Preoperative) to Month 24 (Postoperative)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmHg
Units Other Than Participants: eyes
Arm/Group | XEN® Gel Stent | XEN® Gel Stent With Cataract Surgery
Number analyzed (Participants) | 106 | 79
Number analyzed (eyes) | 114 | 88
mmHg
  Baseline (preoperation) | 21.7 (3.76) | 21.0 (3.39)
  Change from Baseline to Month 24: number analyzed (eyes) | 86 | 75
  Change from Baseline to Month 24 | -6.4 (5.18) | -5.9 (4.60)

4. Primary Outcome: Change From Baseline in the Number of Topical IOP-Lowering Medications in the Study Eyes to Month 24
Description: The use of topical IOP-lowering medications was recorded at the preoperative screening visit and at the 24 Month postoperative visit. The study eye(s) is defined as an eye(s) that met IOP and IOP-lowering medication study inclusion criteria. A negative change from Baseline indicates improvement.
Time Frame: Baseline (≤ 90 days Preoperative) to Month 24 (Postoperative)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: medications
Units Other Than Participants: eyes
Arm/Group | XEN® Gel Stent | XEN® Gel Stent With Cataract Surgery
Number analyzed (Participants) | 106 | 79
Number analyzed (eyes) | 114 | 88
medications
  Baseline (preoperation) | 2.7 (0.93) | 2.5 (0.88)
  Change from Baseline to Month 24: number analyzed (eyes) | 86 | 75
  Change from Baseline to Month 24 | -1.5 (1.54) | -1.5 (1.22)

ADVERSE EVENTS:
Time Frame: Up to 26 Months
Description: The number at risk for Serious Adverse Events and Other Adverse Events (AEs) is based on the number of eyes included in the Safety Population. In this study all AEs were collected at eye level since this is an ophthalmic device. If a participant had both eyes in the study, AEs from each eye were collected separately. Systemic AEs (not local to the participating eyes) were collected twice but to avoid duplication were counted toward the right eyes only.
Arm/Group | XEN® Gel Stent | XEN® Gel Stent With Cataract Surgery
All-Cause Mortality (participants affected / at risk) | 2/112 | 2/87
Serious Adverse Events (participants affected / at risk) | 12/120 | 6/98
Other Adverse Events (participants affected / at risk) | 14/120 | 8/98
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | XEN® Gel Stent (N=120) | XEN® Gel Stent With Cataract Surgery (N=98)
Cardiac arrest (Cardiac disorders) | 1 | 0
Heart attack (Cardiac disorders) | 1 | 0
Cataract aggravated (Eye disorders) | 1 | 0
Retinal disorder (Eye disorders) | 1 | 0
Implant site dehiscence (General disorders) | 0 | 1
Decompensated cirrhosis (Hepatobiliary disorders) | 1 | 0
Endophthalmitis (Infections and infestations) | 1 | 0
Broken hip (Injury, poisoning and procedural complications) | 0 | 2
Intraocular pressure high (Investigations) | 1 | 0
Intraocular pressure high - fellow eye (Investigations) | 0 | 1
Hyponatremia (Metabolism and nutrition disorders) | 1 | 0
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Kidney tumor (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Oral cancer stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Stomach cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Trabeculectomy (Surgical and medical procedures) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | XEN® Gel Stent (N=120) | XEN® Gel Stent With Cataract Surgery (N=98)
Hyphema (Injury, poisoning and procedural complications) | 8 | 2
Trabeculectomy (Surgical and medical procedures) | 7 | 1
YAG (yttrium-aluminum-garnet) laser surgery (Surgical and medical procedures) | 0 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.